CLINICAL TRIAL: NCT07077304
Title: EACVI Study on Multimodality Cardiovascular Imaging of Inflammatory Cardiovascular Diseases
Acronym: EACVI-INFLAME
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: AP-HP250504
Record Dates: First submitted 2025-05-16; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Myocarditis; ANCA Associated Vasculitis; Pericarditis; Systemic Sclerosis; Systemic Lupus Erythematosus; Idiopathic Inflammatory Myopathies; Rheumatoid Arthritis; Spondylarthritis; Behcet Disease; Takayasu Arteritis; Sarcoidosis; Still Disease; Tako Tsubo Cardiomyopathy
Keywords: Cardiovascular disease; Auto-immune disease; Auto-inflammatory disease; Rheumatic disease; CMR; PET; multimodality imaging; ICARD
MeSH Terms: conditions — Myocarditis; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Pericarditis; Scleroderma, Systemic; Lupus Erythematosus, Systemic; Myositis; Arthritis, Rheumatoid; Spondylarthritis; Behcet Syndrome; Takayasu Arteritis; Sarcoidosis; Arthritis, Juvenile; Takotsubo Cardiomyopathy; Cardiovascular Diseases; Rheumatic Diseases | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observational study — observational study

SUMMARY:
Inflammatory Cardiovascular Diseases and Autoimmune Rheumatic Diseases (ICARDs) encompass cardiovascular involvement in connective tissue diseases, vasculitis, and primary inflammatory cardiac processes affecting all layers of the heart. ICARDs are associated with increased cardiovascular morbidity and mortality, independently of traditional risk factors, via multiple pathophysiological mechanisms.

Diagnosis and prognosis are challenged by the heterogeneity of clinical presentations. Multimodality cardiovascular imaging - including cardiovascular magnetic resonance (CMR), transthoracic echocardiography, and positron emission tomography (PET) - plays a central role in detecting and characterizing inflammatory involvement, and may offer prognostic insights.

Given the limited data on the diagnostic and prognostic utility of these imaging modalities in ICARDs, the EACVI-INFLAME study aims to assess the prevalence of confirmed cardiovascular involvement in patients with suspected or established ICARDs undergoing CMR and/or cardiac PET in a multicentric international cohort.

DETAILED DESCRIPTION:
Inflammatory Cardiovascular Diseases and Autoimmune Rheumatic diseases (ICARDs) encompass the cardiovascular manifestations of connective tissue diseases and vasculitis, along with primary inflammation affecting all layers of the heart - such as myocarditis, pericarditis and Tako-Tsubo. ICARDs can result in a vast array of clinical cardiovascular manifestations, including coronary artery disease, acute heart failure, ventricular and supra-ventricular arrhythmia. Autoimmune rheumatic disease have been identified as independent risk factors of major cardiovascular events, even after adjusting for traditional cardiovascular risk factors, and accumulated evidence shows increased cardiovascular morbidity and mortality in ICARDs compared to the general population.

Various pathophysiological mechanisms have been proposed to explain the increased risk of cardiovascular events. Suspected mechanisms include prolonged systemic inflammation, accelerated atherosclerosis, autoantibody and immune complex formation, as well as an increase in sympathetic tone which may contribute to heart failure and arrhythmia. Cardiovascular involvement in patients with ICARDs represents a diagnostic challenge due to the heterogeneity in their clinical presentation, and establishing prognosis following cardiovascular involvement is equally difficult. Multimodality cardiovascular imaging, including cardiovascular magnetic resonance (CMR), transthoracic echocardiography and positron emission tomography (PET) nuclear imaging have emerged as useful diagnostic tools to help differentiate inflammatory diseases among themselves and from other diseases, and identify prognostic markers.

Multimodality cardiovascular imaging has the potential to play a major role in assessing the extent of cardiovascular involvement of both primary inflammatory cardiomyopathies and autoimmune rheumatic diseases, by allowing for an early and more accurate diagnosis, phenotypic classification and monitoring. The additive value of cardiovascular imaging, notably MRI, cardiac PET scan, and multimodality imaging in connective tissue disease and vasculitis remains unclear and has been mentioned as a research topic of interest. Moreover, this study will help acquire data on drug tapering, treatment modalities adapted to different etiologies, as well as data on ICARDs unresponsive to treatment. A thorough assessment of the current practices, diagnostic and prognostic value of multimodality imaging in the context of ICARDs has the potential to help shape future guidelines for early assessment of cardiovascular involvement in ICARDs, and potentially change treatment algorithms.

The establishment of this study is particularly pertinent with the forthcoming ESC guidelines on the management of inflammatory cardiomyopathies, as it will provide real-life data on the application of these guidelines. Due to the lack of evidence in the literature on the topic of the diagnostic and prognostic value of multimodality imaging in the context of ICARDs, this "EACVI-INFLAME" international study will aim to determine the proportion of patients with confirmed cardiovascular involvement in patients with suspected or established ICARDs undergoing CMR and/or cardiac PET in a multicentric international cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Ability to provide informed non-opposition
3. Referred for a CMR and/or nuclear imaging exam

AND a suspicion of one of the following ICARDs :

1. Suspected Myocarditis (acute or chronic, and whatever the aetiologies)
2. Suspected Myocardial Infarction with Non-Obstructive Coronary Arteries (MINOCA)
3. Suspected Tako-Tsubo
4. Suspected Pericarditis (acute or chronic, and whatever the aetiologies)
5. Suspected Connective tissue disease with cardiovascular involvement:

   * Systemic sclerosis
   * Systemic lupus erythematosus
   * Antiphospholipid syndrome
   * Idiopathic inflammatory myopathies
   * Rheumatoid arthritis, spondylarthritis
6. Suspected Vasculitis with cardiovascular involvement:

   * Small-vessel vasculitis (ANCA…)
   * Large vessel vasculitis (Behcet disease, Takayasu…)
7. Suspected Inflammatory disease with cardiovascular involvement:

   * Sarcoidosis
   * Still disease

Exclusion Criteria:

1. Inability to provide non-opposition
2. History of heart transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients with a suspicion of cardiovascular involvement due to a suspected or previously diagnosed ICARD referred for a CMR and/or nuclear imaging exam.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with confirmed cardiovascular involvement among consecutive patients with a suspicion of cardiovascular involvement due to a suspected or known ICARD referred for CMR and/or nuclear imaging exam. | At each diagnostic assessment point, up to study completion, an average of 1 year.
  To assess the proportion of patients with confirmed cardiovascular involvement among consecutive patients with suspected or known ICARD referred for CMR and/or nuclear imaging exam in a multicentre international and prospective study.

SECONDARY OUTCOMES:
Baseline characteristics | At each diagnostic assessment point, up to study completion, an average of 1 year.
  Epidemiologic distribution of clinical, biological and cardiovascular imaging characteristics at baseline.
Proportion of patients presenting with the clinical composite outcome at 1year follow-up | At each diagnostic assessment point, up to study completion, an average of 1 year.
  Proportion of patients presenting with the clinical composite outcome at 1year follow-up defined as the proportion of patients presenting with:
  * Cardiovascular mortality and/or
  * Hospitalization for heart failure (HF) and/or
  * Myocardial infarction and/or
  * Incident atrial fibrillation and/or
  * Stroke and/or
  * Recurrence of ICARD
Proportion of patients with all-cause mortality at 1-year follow-up. | At each diagnostic assessment point, up to study completion, an average of 1 year.
Proportion of patients with cardiovascular mortality at 1-year follow-up. | At each diagnostic assessment point, up to study completion, an average of 1 year.
Proportion of patients hospitalized for heart failure at 1-year follow-up. | At each diagnostic assessment point, up to study completion, an average of 1 year.
Proportion of patients hospitalized for an acute episode of ICARD at 1-year follow-up. | At each diagnostic assessment point, up to study completion, an average of 1 year.
Proportion of patients achieving the remission of ICARD at 1-year follow-up. | At each diagnostic assessment point, up to study completion, an average of 1 year.
Proportion of participants for whom cardiac imaging led to a guideline-concordant diagnosis, according to the cardio-rheumatology team, and specific to each ICARD category. | At each diagnostic assessment point, up to study completion, an average of 1 year.